CLINICAL TRIAL: NCT00454584
Title: A Phase 3, Multicenter, Randomized Study Comparing CNTO 1275 and Etanercept for the Treatment of Moderate to Severe Plaque Psoriasis
Brief Title: An Efficacy and Safety Study of CNTO 1275 Compared to Etanercept in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013015; C0743T12 (Other: Centocor); 2006-003444-30 (EudraCT Number)
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: Psoriasis
Keywords: Psoriasis; CNTO 1275; Etanercept; Immune diorder; Skin disorder
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — Ustekinumab; Etanercept

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CNTO 1275 45 mg (Experimental): Patients will receive CNTO 1275 45 mg at the Weeks 0 and 4 visits. Treatment after Week 12 is dependent on Physician's Global Assessment (PGA) response at Week 12 and initial treatment assignment.
  Interventions: Drug: CNTO 1275 45 mg
- CNTO 1275 90 mg (Experimental): Patients will receive CNTO 1275 90 mg at the Weeks 0 and 4 visits. Treatment after Week 12 is dependent on PGA response at Week 12 and initial treatment assignment.
  Interventions: Drug: CNTO 1275 90 mg
- Etanercept 50 mg (Active Comparator): Patients will receive Etanercept 50 mg twice weekly through Week 12. Treatment after Week 12 is dependent on PGA response at Week 12 and initial treatment assignment.
  Interventions: Drug: Etanercept 50 mg

INTERVENTIONS:
Drug: CNTO 1275 45 mg — Type=exact number, number=45, unit=mg, form=injection, route=subcutaneous
  Arms: CNTO 1275 45 mg
Drug: CNTO 1275 90 mg — Type=exact number, number=90, unit=mg, form=injection, route=subcutaneous
  Arms: CNTO 1275 90 mg
Drug: Etanercept 50 mg — Type=exact number, number=50, unit=mg, form=injection, route=subcutaneous
  Arms: Etanercept 50 mg

SUMMARY:
The purpose of this study is to compare the efficacy and safety of CNTO 1275 to etanercept in patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a multicenter, randomized (study medication assigned by chance), active-controlled, parallel, 3-arm study. Patients will be randomly (allocation to treatments available by chance) assigned in 3:5:5 ratio to receive one of three treatments groups. The three treatment groups are: Group 1 - CNTO 1275 45 mg dosing at weeks 0 and 4, Group 2 - CNTO 1275 90 mg dosing at weeks 0 and 4, Group 3 - Etanercept 50 mg two times per week through week 12. The total duration for each participant will be up to 64 weeks (approximately 16 months). The active-controlled portion of the study is from Week 0 to Week 12 during which the efficacy and safety of etanercept and 2 dose levels of CNTO 1275 will be evaluated. Treatment after Week 12 is dependent on Physician's Global Assessment (PGA) response at Week 12 and initial treatment assignment. Patients will receive 2 subcutaneous injections of CNTO 1275 (either 45 or 90 mg doses) or twice weekly injections of etanercept during the first twelve weeks of the study. Patients may receive two additional doses of CNTO 1275 (either 45 or 90 mg doses) up to week 44.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of plaque-type psoriasis at least 6 months prior to the study
* Have plaque-type psoriasis covering at least 10 percentage of total body surface area
* Have a Psoriasis Area and Severity Index (PASI) score of 12 or greater and a Physician's Global Assessment (PGA) score of 3 or greater at the time of the first administration of study drug
* Must be suitable for phototherapy or systemic treatment for psoriasis
* Have failed to respond to or have condition which prevents use of cyclosporine, methotrexate (MTX) or psoralen plus ultraviolet light A (PUVA)

Exclusion Criteria:

* Currently have nonplaque forms of psoriasis
* Have current drug-induced psoriasis
* Have used any therapeutic agent targeted at reducing interleukin-12 (IL-12) or IL-23 (Interleukins are the substance produced by body in immunological disease like psoriasis)
* Have received phototherapy or any systemic medications/treatments that could affect psoriasis or PASI evaluation (including, but not limited to, oral or injectable corticosteroids, retinoids, 1,25 dihydroxy vitamin D3 and analogues, psoralens, sulfasalazine, hydroxyurea, or fumaric acid derivatives) within 4 weeks of the first administration of study agent
* Have used a biologic within the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Griffiths CE, Strober BE, van de Kerkhof P, Ho V, Fidelus-Gort R, Yeilding N, Guzzo C, Xia Y, Zhou B, Li S, Dooley LT, Goldstein NH, Menter A; ACCEPT Study Group. Comparison of ustekinumab and etanercept for moderate-to-severe psoriasis. N Engl J Med. 2010 Jan 14;362(2):118-28. doi: 10.1056/NEJMoa0810652. PMID 20071701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 903 partcipants received either ustekinumab (CNTO 1275) or etanercept at 67 sites in North America and Europe.
Groups:
- Etanercept (CP): Controlled period (Week 0-12) - Etanercept group
- Ustekinumab 45 mg (CP): Controlled period (Week 0-12) - Ustekinumab 45 mg group
- Ustekinumab 90 mg (CP): Controlled period (Week 0-12) - Ustekinumab 90 mg group
- Etanercept (After CP): After Controlled period (Week 12- 64) - receiving etanercept at Weeks 0 -> receiving ustekinumab 90 mg if becoming a nonresponder during Week 12 and Week 40
- Ustekinumab 45 mg (After CP): After Controlled period (Week 12-64) - receiving ustekinumab 45 mg at Weeks 0 -> retreated with ustekinumab 45 mg if becoming a nonresponder during Week 12 and Week 40.
- Ustekinumab 90 mg (After CP): After Controlled period (Week 12-64) - receiving ustekinumab 90 mg at Weeks 0 -> retreated with ustekinumab 90 mg if becoming a nonresponder during Week 12 and Week 40.
Period: Controlled Period
Arm/Group | Etanercept (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Etanercept (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Started | 347 | 209 | 347 | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.)
Completed | 336 | 201 | 342 | 0 | 0 | 0
Not Completed | 11 | 8 | 5 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 2 | 0 | 0 | 0
Not completed — Other | 5 | 4 | 2 | 0 | 0 | 0
Period: After Controlled Period
Arm/Group | Etanercept (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Etanercept (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Started | 0 ("0" in column indicates this reporting group is not relevant to after Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Controlled Period.) | 336 | 201 | 342
Completed | 0 | 0 | 0 | 310 | 189 | 310
Not Completed | 0 | 0 | 0 | 26 | 12 | 32
Not completed — Adverse Event | 0 | 0 | 0 | 9 | 3 | 9
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 4 | 6
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 13 | 5 | 17

BASELINE CHARACTERISTICS:
Groups:
- Group I: Etanercept: Participants received Etanercept 50 mg twice weekly through Week 12. Participants with PGA greater than or equal to 3 at Week 12 received ustekinumab 90 mg at Week 16 and 20. Participants with PGA leeser than or equal to 2 at Week 12 received ustekinumab 90 mg upon losing PGA response (PGA greater than or equal to 3) and 4 weeks after.
- Group II: Ustekinumab 45 mg: Participants received ustekinumab 45 mg at Weeks 0, 4 . Participants with PGA greater than or equal to 3 at Week 12 received ustekinumab 45 mg at Week 16. Participants with PGA lesser than or equal to 2 at Week 12 received ustekinumab 45 mg upon losing PGA response (PGA greater than or equal to 3) and 4 weeks after.
- Group III: Ustekinumab 90 mg: Participants received ustekinumab 90 mg at Weeks 0, 4 . Participants with PGA greater than or equal to 3 at Week 12 received ustekinumab 90 mg at Week 16. Participants with PGA lesser than or equal to 2 at Week 12 received ustekinumab 90 mg upon losing PGA response (PGA greater than or equal to 3) and 4 weeks after.
- Total: Total of all reporting groups
Arm/Group | Group I: Etanercept | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg | Total
Number analyzed (Participants) | 347 | 209 | 347 | 903
Age Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.40) | 45.1 (12.56) | 44.8 (12.29) | 45.2 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 76 | 113 | 290
  Male | 246 | 133 | 234 | 613

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Greater Than or Equal to 75 Percentage Improvement From Baseline in Psoriasis Area and Severity Index (PASI 75) Score at Week 12
Description: Number of participants achieving greater than or equal to 75 percentage improvement from baseline in Psoriasis Area and Severity Index (PASI) at Week 12. PASI is the widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) -72 (worst). Baseline visit refers to Week 0.
Time Frame: Baseline and Week 12
Population: Intent to treat. All participants randomized were included in the analysis according to the assigned treatment groups. Participants is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy or has missing data at Week 12.
Measure: Number; unit: Participants
Arm/Group | Group I: Etanercept | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg
Number analyzed (Participants) | 347 | 209 | 347
Participants | 197 | 141 | 256
Statistical Analysis 1: Comparison: Group I: Etanercept vs Group III: Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; The test was stratified by baseline weight [<90kg vs. ≥ 90 kg)
Statistical Analysis 2: Comparison: Group I: Etanercept vs Group II: Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 90 mg or 45 mg and etanercept at an overall significant level of 0.05. Sample Size: Assuming the PASI 75 response rates of ustekinumab 90 mg, 45 mg, etanercept are 65%, 64%, and 50% , respectively, with 325 participants each in the ustekinumab 90 mg and etanercept groups, the power to detect a treatment difference is 97%. With 200 participants in the ustekinumab 45 mg group, the complete power to further detect a treatment difference was 87%; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel (CMH) chi square — To control the overall type I error rate at 0.05 level in the primary endpoint analysis, a step-down test procedure was applied. First, ustekinumab 90 mg and etanercept were compared. Then ustekinumab 45 mg and etanercept would be compared; The test was stratified by baseline weight [<90kg vs. ≥ 90 kg)

2. Secondary Outcome: Number of Participants With Physician's Global Assessment (PGA) of Cleared or Minimal at Week 12
Description: Number of participants achieving a physician global assessment (PGA) (0-5) of cleared or minimal at Week 12. The PGA is 7-point scale used in clinical trial of various diseases. In this the physician checks the state of the disease and gives them score from 0 (clear) to 5 (severe).
Time Frame: Week 12
Population: Intent to treat. All randomly assigned participants were included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy or had a missing PGA score.
Measure: Number; unit: Participants
Arm/Group | Group I: Etanercept | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg
Number analyzed (Participants) | 347 | 209 | 347
Participants | 170 | 136 | 245
Statistical Analysis 1: Comparison: Group I: Etanercept vs Group III: Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; The test was stratified by baseline weight [<90kg vs. ≥ 90 kg)
Statistical Analysis 2: Comparison: Group I: Etanercept vs Group II: Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 90 mg or 45 mg and etanercept at an overall significant level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; The test was stratified by baseline weight [<90kg vs. ≥ 90 kg)

3. Secondary Outcome: Number of Participants Achieving a Greater Than or Equal to 90 Percentage Improvement From Baseline in Psoriasis Area and Severity Index (PASI 90) Score at Week 12
Description: Number of participants achieving greater than or equal to 90 percentage improvement from baseline in Psoriasis Area and Severity Index (PASI) at Week 12. PASI is the widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) -72 (worst).
Time Frame: Baseline and Week 12
Population: Intent to treat. All randomly assigned participants were included in the analysis according to the assigned treatment groups. A participant is considered a non-responder if the participant has used any pre-specified prohibited medications, discontinued due to lack of efficacy, or had a missing Week 12 PASI score.
Measure: Number; unit: Participants
Arm/Group | Group I: Etanercept | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg
Number analyzed (Participants) | 347 | 209 | 347
Participants | 80 | 76 | 155
Statistical Analysis 1: Comparison: Group I: Etanercept vs Group III: Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; The test was stratified by baseline weight [<90kg vs. ≥ 90 kg)
Statistical Analysis 2: Comparison: Group I: Etanercept vs Group II: Ustekinumab 45 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; The test was stratified by baseline weight [<90kg vs. ≥ 90 kg)

4. Secondary Outcome: Difference in Psoriasis Area Severity Index Between Week 12 and That Achieved 12 Weeks After Retreatment (Week R12)
Description: The difference between the PASI score at Week 12 and that achieved after 12 weeks of retreatment. The PASI is the widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) -72 (worst).
Time Frame: Up to Week 52. Retreatment may occur anytime between Week 16 and Week 40 depending on time of losing PGA response. Hence end of 12 weeks of retreatment would be between Week 28 and Week 52, inclusive.
Population: Participants who were randomized to ustekinumab, had a PGA score less than or equal to 2 at Week 12, and were retreated upon losing PGA response (PGA greater than or equal to 3).
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg
Number analyzed (Participants) | 152 | 240
Score on a scale | -0.99 (3.799) | -0.30 (4.124)

ADVERSE EVENTS:
Time Frame: Week 64
Description: One participant in Etanercept (after controlled period [CP]), 1 participant in Ustekinumab 90 mg (after CP) and 3 participants stekinumab 45 mg (after CP) arms were discontinued study agent during the CP but had follow-up after CP and hence were included in the tables of frequent adverse events and serious adverse events after CP.
Groups:
- Etanercept (After CP): After Controlled period (Week 12-64) - receiving etanercept at Weeks 0 -> prior to being treated with ustekinumab
- Etanercept -> Ustekinumab 90 mg (After CP): After Controlled period (Week 12-64) - receiving etanercept at Weeks 0 -> receiving ustekinumab 90 mg upon becoming a nonresponder during Week 12 and Week 40. This group is a subpopulation of Etanercept (after CP).
Arm/Group | Etanercept (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Etanercept (After CP) | Etanercept -> Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Serious Adverse Events (participants affected / at risk) | 4/347 | 4/209 | 4/347 | 8/337 | 10/295 | 13/204 | 22/343
Other Adverse Events (participants affected / at risk) | 154/347 | 85/209 | 126/347 | 60/337 | 102/295 | 85/204 | 164/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (CP) (N=347) | Ustekinumab 45 mg (CP) (N=209) | Ustekinumab 90 mg (CP) (N=347) | Etanercept (After CP) (N=337) | Etanercept -> Ustekinumab 90 mg (After CP) (N=295) | Ustekinumab 45 mg (After CP) (N=204) | Ustekinumab 90 mg (After CP) (N=343)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uvulitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Finger amputation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Microangiopathy (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (CP) (N=347) | Ustekinumab 45 mg (CP) (N=209) | Ustekinumab 90 mg (CP) (N=347) | Etanercept (After CP) (N=337) | Etanercept -> Ustekinumab 90 mg (After CP) (N=295) | Ustekinumab 45 mg (After CP) (N=204) | Ustekinumab 90 mg (After CP) (N=343)
Fatigue (General disorders) | 13 | 8 | 19 | 0 | 1 | 5 | 7
Injection site erythema (General disorders) | 53 | 2 | 3 | 0 | 2 | 0 | 5
Injection site haematoma (General disorders) | 25 | 1 | 6 | 0 | 0 | 0 | 2
Injection site swelling (General disorders) | 25 | 3 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 5 | 1 | 4 | 5 | 15 | 10 | 16
Nasopharyngitis (Infections and infestations) | 30 | 21 | 34 | 25 | 38 | 34 | 63
Upper respiratory tract infection (Infections and infestations) | 20 | 13 | 22 | 22 | 35 | 29 | 55
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 11 | 10 | 4 | 7 | 8 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 14 | 15 | 3 | 3 | 5 | 22
Headache (Nervous system disorders) | 38 | 31 | 42 | 5 | 9 | 8 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 5 | 14 | 2 | 3 | 11 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 12 | 16 | 5 | 6 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.